CLINICAL TRIAL: NCT03035006
Title: A Phase I/II, Dose-escalation Study of Lipotecan Based Concurrent Chemoradiotherapy in Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Brief Title: Lipotecan Based Concurrent Chemoradiotherapy in Hepatocellular Carcinoma With Portal Vein Tumor Thrombosis
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Current study design couldn't support futher development on this indication.
Sponsor: Taiwan Liposome Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TLC388A1008
Record Dates: First submitted 2017-01-25; First posted 2017-01-27 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: HepatoCellular Carcinoma; Portal Vein Tumor Thrombosis
Keywords: Hepatocellular carcinoma; Portal vein tumor thrombosis; TLC388; Chemoradiotherapy; Lipotecan
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — TLC 388

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Lipotecan based chemoradiotherapy (Experimental): Patients will receive Lipotecan based CCRT. Lipotecan will be given as a 30-minute (±3 minutes) iv infusion qw for 6 weeks at the predefined dose level for each cohort. A total of 6 doses of Lipotecan will be administered to each patient in conjunction with RT at 3.5 Gy per fraction for 16 fractions. During CCRT period, Lipotecan should be given within 2 hours prior to the start of RT, and the Lipotecan and RT should be delivered on the same day, unless any conditions fulfils with the dose interruption standards. Radiotherapy treatment, at the allocated dose level, is only permitted if the normal tissue dose constrain criteria are maintained
  Interventions: Drug: Lipotecan

INTERVENTIONS:
Drug: Lipotecan — Lipotecan based concurrent chemoradiotherapy
  Other Names: TLC388

SUMMARY:
This is a phase I/II dose-escalation study of lipotecan based concurrent chemoradiotherapy in hepatocellular carcinoma with portal vein tumor thrombosis.

DETAILED DESCRIPTION:
Protocol number: TLCTLC388A1008

Primary objective:

To evaluate the safety and tolerability, including maximum tolerated dose (MTD) and dose-limiting toxicity (DLT), of Lipotecan based concurrent chemoradiotherapy (CCRT) in patients with hepatocellular carcinoma (HCC) and portal vein tumor thrombosis (PVTT) unsuitable for local treatment.

Secondary Objective:

The secondary objective is to explore the efficacy of Lipotecan based CCRT in patients with HCC and PVTT and the effect on quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be males or females

   * ≥20 years of age in Taiwan
   * ≥18 years old in China
2. Patients with histologically confirmed HCC or patients who do not have histological diagnosis, but the lesion is larger than 1 cm in a cirrhotic liver with typical HCC image of contrast enhanced CT scan or MRI. If the image characteristic is not typical of HCC, another contrast enhanced image modality should be confirmed for diagnosis.
3. Patients with PVTT (BCLC stage C) who are not suitable for local therapies
4. Patients with a measureable targeting lesion
5. Patients with an anticipated residual life expectancy ≥3 months
6. Patients who have adequate organ function
7. Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤2
8. Patients who are willing to follow birth control requirements during the study treatment and continue until 2 months after the completion of study treatment
9. Patients willing and able to comply with the study procedures and to sign a written ICF

Exclusion Criteria:

1. Patients with infiltrative type HCC
2. Patients with evidence of any extrahepatic metastasis, including but not limited to inferior vena cava thrombosis, bone metastasis, brain metastasis, or regional lymph node metastasis
3. Patients with a history of West Haven criteria grade III-IV hepatic encephalopathy or ascites
4. Patients with a history of other malignancy except primary HCC within 3 years prior to the screening visit, excluding skin squamous cell carcinoma or basal cell carcinoma
5. Patients who fail to follow the radiation dose constraint in any critical organ in the radiotherapy planning
6. Patients with an inadequately defined hepatic tumor margin for RT planning on MRI or CT that may impact treatment or safety based on investigator's judgment
7. Patients who have experienced significant allergy or hypersensitivity to the contrast medium for CT or MRI that makes it unsafe to perform the delineation for RT planning
8. Patients with a history of liver transplantation
9. Patients with a significant concurrent disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose determination for Lipotecan based CCRT | 3 months
  To determine maximum tolerated dose for Lipotecan based CCRT in HCC patients with portal vein tumor thrombosis
Best objective response evaluation of portal vein tumor thrombosis | 1 year
  To evaluate the best objective response rate of portal vein tumor thrombosis

SECONDARY OUTCOMES:
Conversion rate (CR) of portal vein tumor thrombosis | 1 year
  To evaluate the conversion rate (CR rate) of PVTT
Best overall response of overall disease | 1 year
  To evaluate the best overall response rate of overall disease
Disease control rate of portal vein tumor thrombosis, liver tumors and overall disease | 1 year
  To evaluate DCR of PVTT, liver tumors (target lesions), and overall disease
Time to progression of overall disease | 1 year
  To evaluate the TTP of overall disease after the start of concomitant Lipotecan based CCRT
Progression free survival of overall disease | 1 year
  To evaluate the PFS of overall disease after the start of concomitant Lipotecan based CCRT
Overall survival of overall disease | 1 year
  To evaluate the OS after the start of concomitant Lipotecan based CCRT

CONTACTS AND LOCATIONS:
Overall Officials: Carl Brown, PhD, Study Director — Taiwan Liposome Company
Locations (4):
- Taiwan (4):
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hosipital, Taipei
  - Taipei Veteran General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: Undecided